CLINICAL TRIAL: NCT07396194
Title: Evaluation of the Relation Between Serum Interleukins 17, 38, 41, and HLA-B27 Gene Expression in Ankylosing Spondylitis Patients
Brief Title: Ankylosing Spondylitis
Acronym: Interleukins
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Alaa Ezat Ahmed, Assisstant lecturer, Sohag University
Other Study IDs: Soh-Med-26-1-2MD
Record Dates: First submitted 2026-02-01; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Ankylosing Spondylitis
Keywords: Interleukin 17; Interleukin 38; Interleukin 41; HLA- B27 gene
MeSH Terms: conditions — Spondylitis, Ankylosing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples will be retained
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Patients with Ankylosing spondylitis
- Healthy Controls: Participants Without Ankylosing spondylitis

SUMMARY:
The goal of this observational study is to measure the serum level of cytokines IL-17, IL-38,IL-41, and gene expression of HLA-B27 gene in ankylosing spondylitis patients and healthy control group.

The main question it aims to answer is:

Does the disease activity, severity, serum level of cytokines (IL-17, IL-38, and IL-41) are affected by the HLA-b27 gene positivity?

Researchers will compare the serum level of cytokines IL-17, IL-38,IL-41, and gene expression of HLA-B27 gene in ankylosing spondylitis patients and healthy control group to see if there significant differences in serum levels of interleukins 17, 38, 41 in AS patients and healthy control group.

.

DETAILED DESCRIPTION:
Ankylosing spondylitis (AS) that is known as radiographic SpA (r-axSpA), is a type of axial spondyloarthritis, characterized by the dual pathology of inflammatory bone erosion and aberrant new bone formation. It is characterized by chronic inflammation affecting the sacroiliac joints and spine, leading over time to structural changes such as syndesmophyte formation and spinal ankylosis, with consequent impairment in function and quality of life. As an autoimmune disease, it may also affect several organs, including the eyes, intestines, heart, and lungs .

The global prevalence of AS ranges from 0.3 % to 1.4 %, with a strong predilection for young adult males, in whom mobility and quality of life are often severely impaired. Reports indicate that the global incidence of AS ranges from 0.07 to 0.32%, with a male prevalence 2-3 times higher than that of females .

The etiopathogenesis of spondylo-arthritis is still not fully understood but it has been described as involving several mechanisms of action that synergistically initiate and maintain a pro-inflammatory state, leading to disease onset . Numerous disciplines, including genetics, environment, gut microbiota, and hormones, have previously been studied in relation to the etiology of AS .

Genetic predisposition - particularly carriage of the Human Leukocyte Antigen B27 (HLA-B27) allele - is closely linked to AS susceptibility and underlies several immunopathogenic hallmarks of the disease. There is a growing interest in HLA-B27-based effects, particularly in HLA-B27(+) patients who have AS, although the diagnostic and prognostic functions of HLA-B27 in AS are still being contested. Patients with HLA-B27 positivity have a considerably younger age at onset, a greater number of cases of uveitis, and a higher frequency of involvement of peripheral joints compared to patients with HLA-B27 negative.

The development of inflammatory arthritis is dependent upon the presence of an unbalanced cytokine network. Several interleukins and chemokines, particularly those with pro-inflammatory effects such as tumor necrosis factor (TNF)-α, interleukin (IL)-17A and C-X-C motif chemokine ligand 10 (CXCL10), are involved in mediating inflammation and consequent tissue damage.

IL-17 is a pro-inflammatory cytokine that contributes to the pathogenesis of several inflammatory diseases. The IL-17 family consists of six structurally related cytokines (IL-17A, IL-17B, IL-17C, IL-17D, IL-17E, and IL-17F) . It is a key cytokine which promotes neutrophil recruitment and amplifies Th17 responses. Its serum concentration is also associated with inflammatory activity and response to IL-17 inhibitors.

IL-38 is a recently discovered member of the IL-1 family with anti-inflammatory functions. Functionally, IL-38 is broadly described as a cytokine with anti-inflammatory properties. Pro-inflammatory effects have also been identified and this may depend on IL-38 concentration. Increasing evidence indicates that IL-38 is a vital cytokine in the pathogenesis of several inflammatory autoimmune diseases, such as rheumatoid arthritis (RA), psoriatic arthritis. In AS, although systemic levels of IL-38 have not been determined, an association of IL38 gene polymorphism with AS risk has been proposed.

Metrnl, also referred to as Meteorin-like, Meteorin-b, Subfatin, Cometin, and IL-41, is a novel secretory protein involved in inflammation, immunology, and metabolic regulation that is abundant in organs related to metabolism and barrier tissues. Recent research suggested that Metrnl is involved in bone growth, development, remodeling, and related diseases. The roles of Metrnl in bone formation and resorption remain unclear, so further research is required to establish a clearer link between IL-41 and spinal inflammation in AS patients, which will contribute to understand pathogenesis of AS, and provides a way for the development of practical diagnostic tools and potentially more effective treatments.

The study is a case control study, will be done at Department of Medical Microbiology and Immunology in collaboration with Department of Rheumatology and Rehabilitation, Sohag University Hospitals. The practical part will be done in the Central Research Laboratory, Faculty of Medicine, Sohag University.

-The study will include 84 participants recruited from the outpatient clinics of Rheumatology and Rehabilitation Department, Sohag University Hospitals.

The participants will be divided as follows:

Group 1: 42 patients diagnosed with ankylosing spondylitis who met the 2009 Assessment of Spondyloarthritis International Society (ASAS) classification criteria for axSpA. Disease activity in AS was assessed using the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI).

Patients were stratified into two groups based on BASDAI scores: AS-Stable group (BASDAI ≤ 4) and AS-Active group (BASDAI > 4) Group 2: control group of 42 Age- and sex-matched healthy volunteers who do not suffer from inflammatory or autoimmune diseases belonging to same geographic region.

Aim of the Study:

1. To measure the serum level of cytokines IL-17, IL-38, and IL-41 in ankylosing spondylitis patients (active and stable AS, including patients receiving TNF inhibitors and those not treated by TNF inhibitors) and healthy controls.
2. To measure the gene expression of HLA-b27 gene by qRT-PCR in AS patients and controls.

Methods of the study:

1. Full medical history taking (age, gender, degree of back pain using VAS, morning stiffness duration, and extraarticular manifestations (e.g., uveitis, and psoriasis), family history of AS or any autoimmune diseases, onset, duration of disease, associated diseases, medications, etc). The full patient information page data and consent forms will be completed under the direction of a rheumatologist.
2. Clinical examination with special concern about peripheral, and axial joint examination.
3. Evaluation of AS disease activity by Bath AS disease activity (BASDAI) and Ankylosing Spondylitis Disease Activity Score (ASDAS), functional status by Bath ankylosing spondylitis functional index (BASFI).
4. Comprehensive blood counts (CBC), erythrocyte sedimentation rates (ESR), and C-reactive protein (CRP) .
5. The involvement of the sacroiliac joints will be assessed using the New York criteria.
6. Sacroiliac joints resonance imaging as X rays and MRI.
7. Specimen Collection: Five milliliters of fresh peripheral venous blood will be drawn of study participants and will be placed in tubes containing ethylene-diamine-tetra acetic acid (EDTA).
8. Measuring the serum level of cytokines (IL-17, IL-38, IL-41) will be determined using a commercially available solid-phase enzyme immunoassay kit (ELISA).
9. Measurement of gene expression of HLA-b27 gene in peripheral blood mononuclear cells by qRT-PCR.

Ethical consideration:

-Informed written consent will be obtained from the study group.

ELIGIBILITY:
Inclusion Criteria:

* patients who are diagnosed clinically as ankylosing spondylitis (both active or stable), of either sex , who met the Assessment of Spondyloarthritis International Society (ASAS) criteria for axial spondyloarthritis.

Exclusion Criteria:

* Patients with any autoimmune disorder, chronic illnesses as diabetes mellitus, acute and chronic infectious diseases, malignancy.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be recruited from the outpatient clinics of Rheumatology and Rehabilitation Department, Sohag University Hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
collection of blood samples from paticipants | from March 2026 to August 2026
measurement of serum level of Interleukin 17 in participants | From September 2026 to October 2026
Measurement of serum level of Interleukin 38 in participants | from September 2026 to October 2026
measurement of serum level of Interleukin 41 in participants | from September 2026 to October 2026
measurement of gene expression of HLA- B27 gene in participants | from October 2026 to December 2026

IPD SHARING:
Plan to Share IPD: No
1. to avoid the reuse of data for unfair commercial purposes
  2. to avoid the reuse of data for purposes that had not been approved by participants